CLINICAL TRIAL: NCT01974310
Title: A Randomized Clinical Trial of Face-down Protocol Versus Non-face-down Protocol After Surgery for Macular Holes.
Brief Title: Postoperative Positioning After Surgery for Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Mark Alberti, M.D., Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH-FDP-non-FDP
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Macular Holes
Keywords: Macular Holes; Non face down positioning; Face down positioning
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face-down positioning (Active Comparator): Patients advised face-down positioning after surgery for macular hole.
  Interventions: Procedure: Vitrectomy & Intraocular gas fill; Procedure: Postoperative face-down positioning
- Non-face-down positioning (Experimental): Patients advised non-face-down positioning after surgery for macular hole.
  Interventions: Procedure: Vitrectomy & Intraocular gas fill

INTERVENTIONS:
Procedure: Vitrectomy & Intraocular gas fill
Procedure: Postoperative face-down positioning
  Arms: Face-down positioning

SUMMARY:
Idiopathic macular holes are an important cause of visual loss. Macular holes can be treated by surgically removing the vitreous gel and injecting intraocular gas. Following macular hole surgery, face-down positioning is often advised with the aim of improving the likelihood of macular hole closure. The current evidence of postoperative positioning protocols is insufficient to draw firm conclusions and guide practice. The investigators wish to compare non-face-down positioning and face-down positioning after surgery for macular holes in a randomized trial.

Hypothesis: Non-face-down positioning is equivalent to face-down positioning after surgery for macular holes.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic macular hole stage II-IV
* Informed consent
* Duration of symptoms ≤ 24 months

Exclusion Criteria:

* Previous vitreomacular surgery
* Myopia ≥ 8 diopters
* Ocular trauma
* Disease affecting visual function (proliferative diabetic retinopathy, diabetic macular edema, exudative macular degeneration)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Macular hole closure rate | 3 months
  Macular hole closure rate assessed by optical coherence tomography

SECONDARY OUTCOMES:
ETDRS Visual Acuity Gain | 3 months
Degree of postoperative head incline | 3 days
  Position Sensor
Degree of ocular gas fill | 4 days

OTHER OUTCOMES:
Frequency of the complications | During 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Morten la Cour, Professor, Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, University of Copenhagen, Copenhagen, Denmark